CLINICAL TRIAL: NCT01581359
Title: A Comparative Study, Randomized, Blinded, About the Effect of Pre-treatment With GnRH Analogues Versus Placebo in Infertile Patients With Endometriosis Undergoing in Vitro Fertilization Treatment
Brief Title: The Effect of Pre-treatment With GnRH Analogues Prior in Vitro Fertilization in Patients With Endometriosis
Acronym: ENDOFIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDOFIV-010; 2010-022216-39 (EudraCT Number)
Record Dates: First submitted 2012-03-20; First posted 2012-04-20 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2014-04

CONDITIONS: Endometriosis; Infertility
Keywords: Endometriosis; GnRH treatment; Infertility; IVF
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRHa (Active Comparator): Triptorelin acetate 3,75 mg subcutaneous injection administered on days 1, 28 and 56 after menstrual cycle.
  Interventions: Drug: Triptorelin acetate
- Physiological serum (Placebo Comparator): physiological serum subcutaneous injection with same delivery device and same volume that active comparator ) administered on days 1, 28 and 56 after menstrual cycle.
  Interventions: Drug: Triptorelin acetate

INTERVENTIONS:
Drug: Triptorelin acetate — * Triptorelin acetate Dosing regimen: 1 subcutaneous injection of 3,75 mg/28 days, total of 3 doses
  * Placebo Dosing regimen: subcutaneous injection of the same volume of physiological serum/28 days, total of 3 doses
  Other Names: Gonapeptyl Depot 3,75

SUMMARY:
The purpose of this study is to determine whether the administration of an analogue of gonadotropin-releasing hormone (GnRH) during the three months prior to the performing of an IVF may improve the response to ovarian stimulation, implantation rate and clinical pregnancy rate in patients with endometriosis/ endometriomas.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of ectopic endometrial tissue which induces a local inflammatory reaction. Usually, this tissue is located at any level in the pelvic region, but extrapelvic locations have been described. It is a chronic disease whose cause is unknown, although a genetic predisposition has been proven. It is estimated that endometriosis affects 7-15% of women of fertile age, and up to 30-40% of women with endometriosis have infertility.

Assisted reproduction techniques (ART) are the treatment of many causes of infertility, including endometriosis. The results of assisted reproduction in women with endometriosis appear to be somewhat worse than those obtained from women without endometriosis. Some authors have proven a significant reduction in implantation and pregnancy rates in these patients.

The worst pregnancy rate and implantation is believed to be originated in a poor oocyte quality, which can lead to a lower rate of fertilization. This poor oocyte quality produce poorer quality embryos with a reduced capacity to implant, particularly in severe endometriosis.

On the other hand, endometrial receptivity does not appear to contribute to the reduction of results of ART in these women.

In an attempt to improve ART outcomes in women with endometriosis, different strategies have been proposed prior to the cycle realization, with different results.

Surgical resection of endometriomas (endometriosis cysts) before the cycle of IVF/ICSI may adversely affect the results. On the other hand, careful laparoscopic cystectomy appears not to affect the ovarian response to stimulation.

In addition to surgical approaches, have been tried different medical treatments to improve the results of IVF / intracytoplasmatic sperm injection (ICSI) in women with endometriosis. It has been suggested that treatment with Danazol prior to IVF may improve results. Similarly, prolonged treatment with GnRH analogues few months before IVF could improve the implantation and pregnancy rates. Unfortunately, many of these studies were not randomized and / or controlled so that the true value of therapy with GnRH analogues before IVF in women with endometriosis still needs to be valued. A recent meta-analysis showed that a 3-6 month treatment with GnRH analogues before IVF increased 4 times the odds of clinical pregnancy in women with endometriosis. Nevertheless, these results were concluded from 165 patients and 78 pregnancies, included in 3 clinical trials, which was not specifically to patients with endometriomas.

The lack of studies with proper design, suggests that there is insufficient evidence at present to establish firm recommendations in this regard. This study will contribute to increasing scientific evidence to recommend or not pretreatment with GnRH agonists before IVF en patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with endometriosis diagnosed by surgery in the previous year to their inclusion in the study with signs of residual disease and/or by the existence of ovarian endometrioma in vaginal ecography who are susceptible to IVF treatment.
* BMI < 28 Kg/m2
* Age < 40 years old
* Signed informed consent to perform IVF and participation in this study

Exclusion Criteria:

* Follicle stimulating hormone (FSH) 2nd-5th cycle day > 12 IU/L
* Liver disease (sALAT> 80 IU/L)
* Kidney disease (creatinine > 130 nmol/L)
* Other relevant disease that contraindicates a pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate by started cycle | 2 weeks after biochemical diagnosis of pregnancy
  Number of pregnancies with fetal hearth beat on ultrasound exam divided by total number of started cycle

SECONDARY OUTCOMES:
Number of oocytes retrieved, total and metaphase II | In the moment of oocyte retrieval
Embryo quality | Two-three days after oocyte recovery and IVF
  * A Class: high quality; 4 equal cells, <11% fragmentation, display no irregularities (vacuoles and multinucleation) and normal zona pellucida.
  * B Class: good quality; 2 or 5 cells and <26% fragmentation or 4 cells and 12-25% fragmentation, same or similar size (cells even number), display no irregularities and normal zona pellucida.
  * C Class: intermediate quality; no multinucleation , 3 or 6 cells with <36% fragmentation or 2, 4 and 5 cells with 25-35% fragmentation or inequal size blastomeres or absence/low vacuoles cells or anormal zona pellucida.
Number and size of endometrioma(s) | Day of the Basal ultrasound
  Total number in each ovary, uni or bilateral cysts and maximum diameter (mm) of the biggest endometrioma
Rate of pregnancy to term in patients with endometriosis / endometriomas | 37 weeks after cycle
  Number of deliveries at 37th to 41st weeks of pregnancy divided by total number of pregnancies
Miscarriage rate | 22nd week of pregnancy
  Number of pregnancy losses divided by total number clinical pregnancies
Rate of healthy and live births | 37th to 41st weeks of pregnancy
  Number of healthy and live births divided by total number of started cycle
Fertilization rate | Two days after oocyte recovery and IVF
  Number of cleavage embryos divided by total number of metaphase II oocytes
Total dose of gonadotropins and days of treatment | Day of the administration of human chorionic gonadotropin (hCG)
  Total dose of gonadotropins in IU, and total days on treatment
Cancellation rate and causes | Last day of gonadotropin treatment
  Number of cancelled cycles divided by total number or started cycles
Ovarian Hyperstimulation Syndrome (OHSS) incidence | One month after hCG
  Number of patients diagnosed of OHSS divided by ended cycles. Classification in mild, moderate and severe

CONTACTS AND LOCATIONS:
Overall Officials: ANA Mª MONZÓ, MD, PhD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Human Reproduction Unit of the La Fe University and Politechnic Hospital, Valencia, Valencia, Spain

REFERENCES:
- [Background] Matson PL, Yovich JL. The treatment of infertility associated with endometriosis by in vitro fertilization. Fertil Steril. 1986 Sep;46(3):432-4. doi: 10.1016/s0015-0282(16)49581-6. PMID 3091408
- [Background] Simon C, Gutierrez A, Vidal A, de los Santos MJ, Tarin JJ, Remohi J, Pellicer A. Outcome of patients with endometriosis in assisted reproduction: results from in-vitro fertilization and oocyte donation. Hum Reprod. 1994 Apr;9(4):725-9. doi: 10.1093/oxfordjournals.humrep.a138578. PMID 8046030
- [Background] Arici A, Oral E, Bukulmez O, Duleba A, Olive DL, Jones EE. The effect of endometriosis on implantation: results from the Yale University in vitro fertilization and embryo transfer program. Fertil Steril. 1996 Mar;65(3):603-7. doi: 10.1016/s0015-0282(16)58162-x. PMID 8774295
- [Background] Cahill DJ, Wardle PG, Maile LA, Harlow CR, Hull MG. Ovarian dysfunction in endometriosis-associated and unexplained infertility. J Assist Reprod Genet. 1997 Nov;14(10):554-7. doi: 10.1023/a:1022568331845. PMID 9447453
- [Background] Inoue M, Kobayashi Y, Honda I, Awaji H, Fujii A. The impact of endometriosis on the reproductive outcome of infertile patients. Am J Obstet Gynecol. 1992 Jul;167(1):278-82. doi: 10.1016/s0002-9378(11)91675-5. PMID 1442943
- [Background] Dmowski WP, Rana N, Michalowska J, Friberg J, Papierniak C, el-Roeiy A. The effect of endometriosis, its stage and activity, and of autoantibodies on in vitro fertilization and embryo transfer success rates. Fertil Steril. 1995 Mar;63(3):555-62. doi: 10.1016/s0015-0282(16)57425-1. PMID 7851586
- [Background] Olivennes F, Feldberg D, Liu HC, Cohen J, Moy F, Rosenwaks Z. Endometriosis: a stage by stage analysis--the role of in vitro fertilization. Fertil Steril. 1995 Aug;64(2):392-8. doi: 10.1016/s0015-0282(16)57740-1. PMID 7615119
- [Background] Tanbo T, Omland A, Dale PO, Abyholm T. In vitro fertilization/embryo transfer in unexplained infertility and minimal peritoneal endometriosis. Acta Obstet Gynecol Scand. 1995 Aug;74(7):539-43. doi: 10.3109/00016349509024386. PMID 7618453
- [Background] Huang HY, Lee CL, Lai YM, Chang MY, Chang SY, Soong YK. The outcome of in vitro fertilization and embryo transfer therapy in women with endometriosis failing to conceive after laparoscopic conservative surgery. J Am Assoc Gynecol Laparosc. 1997 May;4(3):299-303. doi: 10.1016/s1074-3804(05)80219-1. PMID 9154777
- [Background] Hickman TN. Impact of endometriosis on implantation. Data from the Wilford Hall Medical Center IVF-ET Program. J Reprod Med. 2002 Oct;47(10):801-8. PMID 12418061
- [Background] Barnhart K, Dunsmoor-Su R, Coutifaris C. Effect of endometriosis on in vitro fertilization. Fertil Steril. 2002 Jun;77(6):1148-55. doi: 10.1016/s0015-0282(02)03112-6. PMID 12057720
- [Background] Wardle PG, Mitchell JD, McLaughlin EA, Ray BD, McDermott A, Hull MG. Endometriosis and ovulatory disorder: reduced fertilisation in vitro compared with tubal and unexplained infertility. Lancet. 1985 Aug 3;2(8449):236-9. doi: 10.1016/s0140-6736(85)90289-2. PMID 2862417
- [Background] Hull MG, Williams JA, Ray B, McLaughlin EA, Akande VA, Ford WC. The contribution of subtle oocyte or sperm dysfunction affecting fertilization in endometriosis-associated or unexplained infertility: a controlled comparison with tubal infertility and use of donor spermatozoa. Hum Reprod. 1998 Jul;13(7):1825-30. doi: 10.1093/humrep/13.7.1825. PMID 9740433
- [Background] Bergendal A, Naffah S, Nagy C, Bergqvist A, Sjoblom P, Hillensjo T. Outcome of IVF in patients with endometriosis in comparison with tubal-factor infertility. J Assist Reprod Genet. 1998 Oct;15(9):530-4. doi: 10.1023/a:1022526002421. PMID 9822979
- [Background] Pal L, Shifren JL, Isaacson KB, Chang Y, Leykin L, Toth TL. Impact of varying stages of endometriosis on the outcome of in vitro fertilization-embryo transfer. J Assist Reprod Genet. 1998 Jan;15(1):27-31. doi: 10.1023/a:1022574221115. PMID 9493063
- [Background] Norenstedt SN, Linderoth-Nagy C, Bergendal A, Sjoblom P, Bergqvist A. Reduced developmental potential in oocytes from women with endometriosis. J Assist Reprod Genet. 2001 Dec;18(12):644-9. doi: 10.1023/a:1013111200251. PMID 11808845
- [Background] O'Shea RT, Chen C, Weiss T, Jones WR. Endometriosis and in-vitro fertilisation. Lancet. 1985 Sep 28;2(8457):723. doi: 10.1016/s0140-6736(85)92957-5. No abstract available. PMID 2863700
- [Background] Yovich JL, Yovich JM, Tuvik AI, Matson PL, Willcox DL. In-vitro fertilisation for endometriosis. Lancet. 1985 Sep 7;2(8454):552. doi: 10.1016/s0140-6736(85)90485-4. No abstract available. PMID 2863565
- [Background] Garrido N, Navarro J, Remohi J, Simon C, Pellicer A. Follicular hormonal environment and embryo quality in women with endometriosis. Hum Reprod Update. 2000 Jan-Feb;6(1):67-74. doi: 10.1093/humupd/6.1.67. PMID 10711831
- [Background] Pellicer A, Valbuena D, Bauset C, Albert C, Bonilla-Musoles F, Remohi J, Simon C. The follicular endocrine environment in stimulated cycles of women with endometriosis: steroid levels and embryo quality. Fertil Steril. 1998 Jun;69(6):1135-41. doi: 10.1016/s0015-0282(98)00085-5. PMID 9627305
- [Background] Pellicer A, Albert C, Mercader A, Bonilla-Musoles F, Remohi J, Simon C. The follicular and endocrine environment in women with endometriosis: local and systemic cytokine production. Fertil Steril. 1998 Sep;70(3):425-31. doi: 10.1016/s0015-0282(98)00204-0. PMID 9757870
- [Background] Smith MP, Keay SD, Margo FC, Harlow CR, Wood PJ, Cahill DJ, Hull MG. Total cortisol levels are reduced in the periovulatory follicle of infertile women with minimal-mild endometriosis. Am J Reprod Immunol. 2002 Jan;47(1):52-6. doi: 10.1034/j.1600-0897.2002.1o122.x. PMID 11885559
- [Background] Cunha-Filho JS, Lemos NA, Freitas FM, Kiefer K, Faller M, Passos EP. Insulin-like growth factor (IGF)-1 and IGF binding protein-1 and -3 in the follicular fluid of infertile patients with endometriosis. Hum Reprod. 2003 Feb;18(2):423-8. doi: 10.1093/humrep/deg077. PMID 12571183
- [Background] Carlberg M, Nejaty J, Froysa B, Guan Y, Soder O, Bergqvist A. Elevated expression of tumour necrosis factor alpha in cultured granulosa cells from women with endometriosis. Hum Reprod. 2000 Jun;15(6):1250-5. doi: 10.1093/humrep/15.6.1250. PMID 10831550
- [Background] Nakahara K, Saito H, Saito T, Ito M, Ohta N, Takahashi T, Hiroi M. Ovarian fecundity in patients with endometriosis can be estimated by the incidence of apoptotic bodies. Fertil Steril. 1998 May;69(5):931-5. doi: 10.1016/s0015-0282(98)00038-7. PMID 9591505
- [Background] Toya M, Saito H, Ohta N, Saito T, Kaneko T, Hiroi M. Moderate and severe endometriosis is associated with alterations in the cell cycle of granulosa cells in patients undergoing in vitro fertilization and embryo transfer. Fertil Steril. 2000 Feb;73(2):344-50. doi: 10.1016/s0015-0282(99)00507-5. PMID 10685541
- [Background] Sung L, Mukherjee T, Takeshige T, Bustillo M, Copperman AB. Endometriosis is not detrimental to embryo implantation in oocyte recipients. J Assist Reprod Genet. 1997 Mar;14(3):152-6. doi: 10.1007/BF02766132. PMID 9090558
- [Background] Pellicer A, Oliveira N, Ruiz A, Remohi J, Simon C. Exploring the mechanism(s) of endometriosis-related infertility: an analysis of embryo development and implantation in assisted reproduction. Hum Reprod. 1995 Dec;10 Suppl 2:91-7. doi: 10.1093/humrep/10.suppl_2.91. PMID 8745306
- [Background] Ho HY, Lee RK, Hwu YM, Lin MH, Su JT, Tsai YC. Poor response of ovaries with endometrioma previously treated with cystectomy to controlled ovarian hyperstimulation. J Assist Reprod Genet. 2002 Nov;19(11):507-11. doi: 10.1023/a:1020970417778. PMID 12484492
- [Background] Aboulghar MA, Mansour RT, Serour GI, Al-Inany HG, Aboulghar MM. The outcome of in vitro fertilization in advanced endometriosis with previous surgery: a case-controlled study. Am J Obstet Gynecol. 2003 Feb;188(2):371-5. doi: 10.1067/mob.2003.13. PMID 12592242
- [Background] Canis M, Pouly JL, Tamburro S, Mage G, Wattiez A, Bruhat MA. Ovarian response during IVF-embryo transfer cycles after laparoscopic ovarian cystectomy for endometriotic cysts of >3 cm in diameter. Hum Reprod. 2001 Dec;16(12):2583-6. doi: 10.1093/humrep/16.12.2583. PMID 11726578
- [Background] Marconi G, Vilela M, Quintana R, Sueldo C. Laparoscopic ovarian cystectomy of endometriomas does not affect the ovarian response to gonadotropin stimulation. Fertil Steril. 2002 Oct;78(4):876-8. doi: 10.1016/s0015-0282(02)03326-5. PMID 12372472
- [Background] Donnez J, Wyns C, Nisolle M. Does ovarian surgery for endometriomas impair the ovarian response to gonadotropin? Fertil Steril. 2001 Oct;76(4):662-5. doi: 10.1016/s0015-0282(01)02011-8. PMID 11591395
- [Background] Wyns C, Donnez J. [Laser vaporization of ovarian endometriomas: the impact on the response to gonadotrophin stimulation]. Gynecol Obstet Fertil. 2003 Apr;31(4):337-42. doi: 10.1016/s1297-9589(03)00069-9. French. PMID 12821063
- [Background] Garcia-Velasco JA, Mahutte NG, Corona J, Zuniga V, Giles J, Arici A, Pellicer A. Removal of endometriomas before in vitro fertilization does not improve fertility outcomes: a matched, case-control study. Fertil Steril. 2004 May;81(5):1194-7. doi: 10.1016/j.fertnstert.2003.04.006. PMID 15136074
- [Background] Dicker D, Goldman JA, Feldberg D, Ashkenazi J, Levy T. Transvaginal ultrasonic needle-guided aspiration of endometriotic cysts before ovulation induction for in vitro fertilization. J In Vitro Fert Embryo Transf. 1991 Oct;8(5):286-9. doi: 10.1007/BF01139786. PMID 1757743
- [Background] Suganuma N, Wakahara Y, Ishida D, Asano M, Kitagawa T, Katsumata Y, Moriwaki T, Furuhashi M. Pretreatment for ovarian endometrial cyst before in vitro fertilization. Gynecol Obstet Invest. 2002;54 Suppl 1:36-40; discussion 41-2. doi: 10.1159/000066293. PMID 12441659
- [Background] Dicker D, Ashkenazi J, Feldberg D, Levy T, Dekel A, Ben-Rafael Z. Severe abdominal complications after transvaginal ultrasonographically guided retrieval of oocytes for in vitro fertilization and embryo transfer. Fertil Steril. 1993 Jun;59(6):1313-5. doi: 10.1016/s0015-0282(16)55997-4. PMID 8495784
- [Background] Yaron Y, Peyser MR, Samuel D, Amit A, Lessing JB. Infected endometriotic cysts secondary to oocyte aspiration for in-vitro fertilization. Hum Reprod. 1994 Sep;9(9):1759-60. doi: 10.1093/oxfordjournals.humrep.a138789. PMID 7836533
- [Background] Nargund G, Parsons J. Infected endometriotic cysts secondary to oocyte aspiration for in-vitro fertilization. Hum Reprod. 1995 Jun;10(6):1555. doi: 10.1093/humrep/10.6.1555-a. No abstract available. PMID 7593536
- [Background] Younis JS, Ezra Y, Laufer N, Ohel G. Late manifestation of pelvic abscess following oocyte retrieval, for in vitro fertilization, in patients with severe endometriosis and ovarian endometriomata. J Assist Reprod Genet. 1997 Jul;14(6):343-6. doi: 10.1007/BF02765839. PMID 9226514
- [Background] Wei CF, Chen SC. Pelvic abscess after ultrasound-guided aspiration of endometrioma: a case report. Zhonghua Yi Xue Za Zhi (Taipei). 1998 Oct;61(10):603-7. PMID 9830238
- [Background] Kim CH, Chae HD, Kang BM, Chang YS, Mok JE. The immunotherapy during in vitro fertilization and embryo transfer cycles in infertile patients with endometriosis. J Obstet Gynaecol Res. 1997 Oct;23(5):463-70. doi: 10.1111/j.1447-0756.1997.tb00874.x. PMID 9392913
- [Background] Tei C, Miyazaki T, Kuji N, Tanaka M, Sueoka K, Yoshimura Y. Effect of danazol on the pregnancy rate in patients with unsuccessful in vitro fertilization-embryo transfer. J Reprod Med. 1998 Jun;43(6):541-6. PMID 9653702
- [Background] Oehninger S, Brzyski RG, Muasher SJ, Acosta AA, Jones GS. In-vitro fertilization and embryo transfer in patients with endometriosis: impact of a gonadotrophin releasing hormone agonist. Hum Reprod. 1989 Jul;4(5):541-4. doi: 10.1093/oxfordjournals.humrep.a136941. PMID 2507576
- [Background] Dicker D, Goldman GA, Ashkenazi J, Feldberg D, Voliovitz I, Goldman JA. The value of pre-treatment with gonadotrophin releasing hormone (GnRH) analogue in IVF-ET therapy of severe endometriosis. Hum Reprod. 1990 May;5(4):418-20. doi: 10.1093/oxfordjournals.humrep.a137114. PMID 2113929
- [Background] Dale PO, Tanbo T, Abyholm T. Endometriosis-associated infertility treated by long-term gonadotropin-releasing hormone agonist administration and assisted fertilization. J In Vitro Fert Embryo Transf. 1990 Jun;7(3):180-1. doi: 10.1007/BF01135686. PMID 2116489
- [Background] Nakamura K, Oosawa M, Kondou I, Inagaki S, Shibata H, Narita O, Suganuma N, Tomoda Y. Menotropin stimulation after prolonged gonadotropin releasing hormone agonist pretreatment for in vitro fertilization in patients with endometriosis. J Assist Reprod Genet. 1992 Apr;9(2):113-7. doi: 10.1007/BF01203749. PMID 1627925
- [Background] Curtis P, Jackson A, Bernard A, Shaw RW. Pretreatment with gonadotrophin releasing hormone (GnRH) analogue prior to in vitro fertilisation for patients with endometriosis. Eur J Obstet Gynecol Reprod Biol. 1993 Dec 30;52(3):211-6. doi: 10.1016/0028-2243(93)90074-m. PMID 8163038
- [Background] Marcus SF, Edwards RG. High rates of pregnancy after long-term down-regulation of women with severe endometriosis. Am J Obstet Gynecol. 1994 Sep;171(3):812-7. doi: 10.1016/0002-9378(94)90103-1. PMID 8092234
- [Background] Chedid S, Camus M, Smitz J, Van Steirteghem AC, Devroey P. Comparison among different ovarian stimulation regimens for assisted procreation procedures in patients with endometriosis. Hum Reprod. 1995 Sep;10(9):2406-11. doi: 10.1093/oxfordjournals.humrep.a136308. PMID 8530675
- [Background] Ruiz-Velasco V, Allende S. Goserelin followed by assisted reproduction: results in infertile women with endometriosis. Int J Fertil Womens Med. 1998 Jan-Feb;43(1):18-23. PMID 9532465
- [Background] Sallam HN, Garcia-Velasco JA, Dias S, Arici A. Long-term pituitary down-regulation before in vitro fertilization (IVF) for women with endometriosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004635. doi: 10.1002/14651858.CD004635.pub2. PMID 16437491